CLINICAL TRIAL: NCT03759392
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Assess the Effect of Omecamtiv Mecarbil on Exercise Capacity in Subjects With Heart Failure With Reduced Ejection Fraction and Decreased Exercise Tolerance
Brief Title: Study to Assess the Effect of Omecamtiv Mecarbil on Exercise Capacity in Subjects With Heart Failure
Acronym: METEORIC-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 1031; 2018-001233-40 (EudraCT Number)
Record Dates: First submitted 2018-11-15; First posted 2018-11-30 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — omecamtiv mecarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omecamtiv Mecarbil (Experimental): Omecamtiv mecarbil was administered as an oral modified-release tablet twice daily for up to 20 weeks. Participants randomized to this arm started at an omecamtiv mecarbil dose of 25 mg twice daily. The dose could be increased based on plasma concentrations at Weeks 2 and 6.
  Interventions: Drug: Omecamtiv Mecarbil
- Placebo (Placebo Comparator): Participants randomized this arm received placebo tablets (matching the appearance of the omecamtiv mecarbil tablets) twice daily for up to 20 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omecamtiv Mecarbil — Oral omecamtiv mecarbil twice daily for up to 20 weeks with dose level determined by periodic blood testing
  Other Names: CK-1827452; AMG-423
  Arms: Omecamtiv Mecarbil
Drug: Placebo — Oral placebo twice daily for up to 20 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of treatment with omecamtiv mecarbil compared with placebo on exercise capacity as determined by cardiopulmonary exercise testing following 20 weeks of treatment with omecamtiv mecarbil or placebo

DETAILED DESCRIPTION:
Oversight Authorities:

United States: Food and Drug Administration Canada: Health Canada France: National Agency for the Safety of Medicine and Health Products Germany: Federal Institute for Drugs and Medical Devices Hungary: National Institute of Pharmacy and Nutrition Italy: Italian Medicines Agency Netherlands: Medicines Evaluation Board Poland: Chief Pharmaceutical Inspectorate Sweden: Medical Products Agency

ELIGIBILITY:
Inclusion Criteria

* Male or female, greater than or equal to 18 to lesser than or equal to 85 years of age
* History of chronic HF, defined as requiring continuous treatment with medications for HF for a minimum of 3 months before screening
* New York Heart Association (NYHA) class II or III at screening
* Left ventricular ejection fraction less than or equal to 35%
* On maximally tolerated HF standard of care (SoC) therapies consistent with regional clinical practice guidelines, if not contraindicated and according to investigator judgment of the subject's clinical status. Beta blocker dose must be stable for 30 days prior to randomization.
* N-terminal (NT)-proBNP level greater than or equal to 200 pg/mL
* Peak VO2 less than or equal to 75% of the predicted normal value with respiratory exchange ratio (RER) greater than or equal to 1.05 on a screening CPET, confirmed by a CPET core laboratory

Exclusion Criteria

* Severe uncorrected valvular heart disease
* Paroxysmal atrial fibrillation or flutter documented within the previous 6 months, direct-current (DC) cardioversion or ablation procedure for atrial fibrillation within 6 months, or plan to attempt to restore sinus rhythm within 6 months of randomization. Subjects with persistent atrial fibrillation and no sinus rhythm documented in the prior 6 months are permitted.
* Symptomatic bradycardia, second-degree Mobitz type II, or third-degree heart block without a pacemaker.
* History of gastrointestinal bleeding requiring hospitalization, urgent procedure or transfusion in the prior year, or received intravenous (IV) iron, blood transfusion, or an erythropoiesis-stimulating agent (ESA) within 3 months prior to screening, or planned blood transfusion or ESA use during the study screening or treatment period. Chronic, stable use of oral iron is permitted.
* Ongoing or planned enrollment in cardiac rehabilitation.
* Requires assistance to walk or use of mobility assistive devices such as motorized devices, wheelchairs, or walkers. The use of canes for stability while ambulating is acceptable if the subject is deemed capable of performing CPET.
* Major medical event or procedure within 3 months prior to randomization, including: hospitalization, surgery, renal replacement therapy or cardiac procedure. This includes episodes of decompensated HF that require IV HF treatment.
* At screening: Resting systolic BP greater than 140 mmHg or less than 85 mmHg, or diastolic BP greater than 90 mmHg (mean of triplicate readings); Resting heart rate greater than 90 beats per minute, or less than 50 beats per minute (mean of triplicate readings); Estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73m2 (by the modified Modification of Diet in Renal Disease equation); Hepatic impairment defined by a total bilirubin (TBL) greater than or equal to 2 times the upper limit of normal (ULN), or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than or equal to 3 times ULN. Patients with documented Gilbert syndrome and TBL greater than or equal to 2 times ULN due to unconjugated hyperbilirubinemia, without other hepatic impairment, are permitted.
* Room air oxygen saturation under 90% at screening
* Hemoglobin less than 10.0 g/dL at screening
* Significant adverse finding (e.g., exercise-induced early ischemic changes, abnormal decrease in BP [systolic BP falls by more than 10 mmHg], unexpected arrhythmia or other serious finding) during CPET at screening that precludes safe participation in the study, per investigator
* Chronotropic incompetence (including inadequate pacemaker rate response) during CPET at screening, defined as a maximum heart rate <60% of the maximum predicted heart rate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2022-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics, MD, Study Director — Cytokinetics
Locations (81):
- United States (36):
  - Alaska Heart and Vascular Institute, Anchorage, Alaska
  - Arkansas Cardiology Clinic, Little Rock, Arkansas
  - Harbor-UCLA Medical Center, Torrance, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Hartford Hospital-University of Connecticut School of Medicine, Hartford, Connecticut
  - Holy Cross Hospital - Fort Lauderdale, Fort Lauderdale, Florida
  - Broward Research Center - Pembroke Pines, Pembroke Pines, Florida
  - Emory University, Atlanta, Georgia
  - Community Hospital South, Inc., Indianapolis, Indiana
  - Saint Vincent Medical Group Inc., Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital (MGH) - Cardiac Unit Associates, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Heart & Vascular Institute, Detroit, Michigan
  - McLaren Health Care Corporation, Petoskey, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Saint Luke's Health System, Kansas City, Missouri
  - Glacier View Research Institute, Cardiology, Kalispell, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cardiovascular Associates Of The Delaware Valley (Cadv), P.A. - Elmer Physicians Care Center - Elmer, Elmer, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Queens Heart Institute, Rosedale, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Med Health and Hospital, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - St. John Clinical Research Institute, Tulsa, Oklahoma
  - Oregon Health, Portland, Oregon
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Lancaster Heart And Stroke Foundation, Lancaster, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - University of Texas - Southwestern Medical Center, Dallas, Texas
  - Baylor Scott and White Heart and Vascular Hospital, Dallas, Texas
  - Inova Heart and Vascular Institute, Falls Church, Virginia
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Universite de Montreal Institut de Cardiologie de Montreal ICM Montreal Heart Institute MHI, Montreal, Quebec
  - Mcgill University Health Centre (MUHC)-The Montreal General Hospital (MGH), Montreal, Quebec
- France (7):
  - Centre Hospitalier De La Cote Basque, Bayonne
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Centre Hospitalier Universitaire de Grenoble-Hopital Albert Michallon, La Tronche
  - Universite De Nantes - L'Institut Du Thorax, Nantes
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Lariboisiere, Paris
  - Chu de Rouen Hopital Charles Nicolle, Rouen
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hopital Rangueil, Toulouse
- Germany (6):
  - Universitaetsklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - Universitaetsklinikum Jena, Jena, Thuringia
  - Kerckhoff-Klinik- Bad Nauheim, Bad Nauheim
  - Praxisklinik Dresden, Dresden
  - Universitaetsklinikum Des Saarlandes Und Medizinische Fakultaet Der Universitaet Des Saarlandes, Homburg
- Hungary (3):
  - Balatonfuredi Allami Szivkorhaz, Balatonfüred
  - Semmelweis University Heart and Vascular Center, Budapest
  - Pecsi Tudomanyegyetem (PTE) Altalanos Orvostudomanyi Kar (AOK) (University of Pecs Medical School), Pécs
- Italy (7):
  - Ospedali Riuniti Foggia, Foggia, Apulia
  - Centro Cardiologico Monzino IRCCS, Milan, Lombardy
  - Azienda Ospedaliera S.Orsola Malpighi, Bologna, Province of Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia, Province Of Brescia
  - Insituto Di Ricovero E Cura A Carattere Scientifico San Raffaele Pisana, Roma, Rome
  - Divisione di Cardiologia con Utic ed Emodinamica, Napoli
  - Ospedale Monaldi, Napoli
- Netherlands (8):
  - Erasmus MC - Universitair Medisch Centrum Rotterdam, Rotterdam, South Holland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis (OLVG) Locatie West, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Radboud Universiteit - Radboud Universitair Medisch Centrum (Radboudumc), Nijmegen
  - Universitair Medisch Centrum Utrecht - Wilhelmina Kinderziekenhuis, Utrecht
  - Maxima Medisch Centrum Veldhoven, Veldhoven
- Poland (7):
  - Centrum Medyczne Medyk Sp z o.o. Sp. k., Rzeszów, Podkarpackie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Uniwersyteckie Centrum Kliniczne Kliniczne Centrum Kardiologii, Gdansk
  - Oddzial Kliniczny Choroby Wiencowej i Niewydolnosci Serca z Pododdzialem Intensywnego Nadzoru Kardiologicznego, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika, Oddzial Kardiologiczny, Lodz
  - Instytut Kardiologii Heart Failure Clinic, Warsaw
  - Centrum Chorob Serca, Uniwersytecki Szpital Kllniczny im. Jana Mikulicza Radeckiego we Wrociawiu, Wroclaw
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Enhet Klinisk forskning, hjartmedicin, Skanes Universitet Sjukhus, Lund

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Lewis GD, Voors AA, Cohen-Solal A, Metra M, Whellan DJ, Ezekowitz JA, Bohm M, Teerlink JR, Docherty KF, Lopes RD, Divanji PH, Heitner SB, Kupfer S, Malik FI, Meng L, Wohltman A, Felker GM. Effect of Omecamtiv Mecarbil on Exercise Capacity in Chronic Heart Failure With Reduced Ejection Fraction: The METEORIC-HF Randomized Clinical Trial. JAMA. 2022 Jul 19;328(3):259-269. doi: 10.1001/jama.2022.11016. PMID 35852527
- [Derived] Lewis GD, Docherty KF, Voors AA, Cohen-Solal A, Metra M, Whellan DJ, Ezekowitz JA, Ponikowski P, Bohm M, Teerlink JR, Heitner SB, Kupfer S, Malik FI, Meng L, Felker GM. Developments in Exercise Capacity Assessment in Heart Failure Clinical Trials and the Rationale for the Design of METEORIC-HF. Circ Heart Fail. 2022 May;15(5):e008970. doi: 10.1161/CIRCHEARTFAILURE.121.008970. Epub 2022 Mar 3. PMID 35236099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with heart failure with reduced ejection fraction (HFrEF) were enrolled at 63 sites in Canada, France, Germany, Hungary, Italy, Netherlands, Poland, Sweden, and the United States. The first participant enrolled on 09 April 2019, and the last participant completed follow-up on 06 January 2022.
Pre-assignment Details: A total of 276 participants were randomized in a 2:1 ratio to treatment: 185 to omecamtiv mecarbil and 91 to placebo.
Groups:
- Omecamtiv Mecarbil: Omecamtiv mecarbil was administered as an oral modified release tablet twice daily for up to 20 weeks. Participants randomized to this arm started at an omecamtiv mecarbil dose of 25 mg twice daily. The dose could be increased based on plasma concentrations at Weeks 2 and 6.
- Placebo: Participants randomized to this arm received placebo tablets (matching the appearance of the omecamtiv mecarbil tablets) twice daily for up to 20 weeks.
Period: Overall Study
Arm/Group | Omecamtiv Mecarbil | Placebo
Started | 185 | 91
Completed | 164 | 85
Not Completed | 21 | 6
Not completed — Adverse Event | 12 | 4
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Consistently forgot to bring study drug kits to site visits (for compliance check) | 1 | 0
Not completed — No longer able to take medicines | 1 | 0
Not completed — Stopped taking study drug | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omecamtiv Mecarbil | Placebo | Total
Number analyzed (Participants) | 185 | 91 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.64) | 64.4 (11.41) | 63.6 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 15 | 42
  Male | 158 | 76 | 234
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 6 | 22
  White | 163 | 82 | 245
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Time since HFrEF diagnosis [Mean (Standard Deviation); unit: years] — Population: The time since HFrEF diagnosis was missing for 1 participant in the omecamtiv mecarbil arm.
  years
    number analyzed (Participants) | 184 | 91 | 275
    (all) | 7.6 (6.14) | 7.8 (6.88) | 7.7 (6.38)
Primary cause of heart failure: ischemic heart disease [Count of Participants; unit: Participants] | 117 | 48 | 165

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Oxygen Uptake on Cardiopulmonary Exercise Testing From Baseline to Week 20
Description: The effect of treatment on exercise capacity, as assessed by peak oxygen uptake, was assessed during cardiopulmonary exercise testing (CPET) with gas-exchange analysis. Cycle ergometry was the preferred modality for exercise testing; treadmill exercise testing was an acceptable alternative. Participants were to use the same testing modality for all exercise tests during the study. Whenever possible, CPET was administered by the same study personnel using the same equipment throughout the study.
Time Frame: Baseline and Week 20
Population: Full Analysis Set (all randomized participants who received at least 1 dose of randomized study drug)
Measure: Least Squares Mean (Standard Error); unit: mL/min/kg
Arm/Group | Omecamtiv Mecarbil | Placebo
Number analyzed (Participants) | 162 | 81
mL/min/kg | -0.239 (0.1718) | 0.207 (0.2412)
Statistical Analysis 1: Comparison: Omecamtiv Mecarbil vs Placebo; Test type: Superiority; p = 0.13, ANCOVA; Using multiple imputation; Least squares mean difference = -0.447, 95% CI 2-sided [-1.024 to 0.131], Standard Error of Mean 0.2931

2. Secondary Outcome: Change in Total Workload During Cardiopulmonary Exercise Testing From Baseline to Week 20
Description: Total workload was measured during CPET (cycle ergometry [preferred] or treadmill exercise testing) and represents the maximum load to which a participant was subjected during CPET in order to produce work.
Time Frame: Baseline and Week 20
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Watt
Arm/Group | Omecamtiv Mecarbil | Placebo
Number analyzed (Participants) | 162 | 81
Watt | -3.798 (1.3352) | 1.590 (1.9477)
Statistical Analysis 1: Comparison: Omecamtiv Mecarbil vs Placebo; Test type: Superiority; p = 0.025, ANCOVA; Using multiple imputation; Least squares mean difference = -5.388, 95% CI 2-sided [-10.108 to -0.0668], Standard Error of Mean 2.3937

3. Secondary Outcome: Change in Ventilatory Efficiency During Cardiopulmonary Exercise Testing From Baseline to Week 20
Description: Ventilatory efficiency (ventilation [VE]/volume of exhaled carbon dioxide [VCO2]) was measured through CPET with gas exchange analysis.
Time Frame: Baseline and Week 20
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: slope
Arm/Group | Omecamtiv Mecarbil | Placebo
Number analyzed (Participants) | 162 | 81
slope | 0.277 (0.3616) | -0.138 (0.5065)
Statistical Analysis 1: Comparison: Omecamtiv Mecarbil vs Placebo; Test type: Superiority; p = 0.51, ANCOVA; Using multiple imputation; Least squares mean difference = 0.414, 95% CI 2-sided [-0.810 to 1.639], Standard Error of Mean 0.6215

4. Secondary Outcome: Change in the Average Daily Activity Units Measured Over a 2-week Period From Baseline (Week -2 to Day 1) to Weeks 18-20
Description: The effect of treatment on daily activity, as assessed by average daily activity units, was evaluated by actigraphy. Actigraphy was collected during 4 sessions throughout the study for 2 week intervals.
Time Frame: Baseline (Week -2 to Day 1) to Weeks 18-20
Population: The analysis population included participants in the Full Analysis Set with available data at both assessment time frames (ie, baseline [Week -2 to Day 1] and Weeks 18-20).
Measure: Least Squares Mean (Standard Error); unit: 10^5 activity units
Arm/Group | Omecamtiv Mecarbil | Placebo
Number analyzed (Participants) | 147 | 77
10^5 activity units | -0.2 (0.30) | -0.5 (0.38)
Statistical Analysis 1: Comparison: Omecamtiv Mecarbil vs Placebo; Test type: Superiority; p = 0.54, Repeated measures mixed model; Least squares mean difference = 0.3, 95% CI 2-sided [-0.6 to 1.1], Standard Error of Mean 0.42

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization through the end of study/safety follow-up visit (scheduled to occur 4 weeks after the last dose of study drug) or 30 days after the last dose of study drug, whichever was later.
Arm/Group | Omecamtiv Mecarbil | Placebo
All-Cause Mortality (participants affected / at risk) | 3/185 | 1/91
Serious Adverse Events (participants affected / at risk) | 30/185 | 13/91
Other Adverse Events (participants affected / at risk) | 126/185 | 58/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omecamtiv Mecarbil (N=185) | Placebo (N=91)
Cardiac failure (Cardiac disorders) | 7 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 5 | 2
Cardiac arrest (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Hypotension (Vascular disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplanted heart (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Heart transplant (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omecamtiv Mecarbil (N=185) | Placebo (N=91)
Cardiac failure (Cardiac disorders) | 5 | 2
Angina pectoris (Cardiac disorders) | 4 | 3
Atrial fibrillation (Cardiac disorders) | 4 | 3
Palpitations (Cardiac disorders) | 0 | 2
Fatigue (General disorders) | 9 | 4
Non-cardiac chest pain (General disorders) | 4 | 3
Asthenia (General disorders) | 4 | 0
Chest discomfort (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Nausea (Gastrointestinal disorders) | 3 | 3
Fall (Injury, poisoning and procedural complications) | 7 | 1
Dizziness (Nervous system disorders) | 9 | 5
Headache (Nervous system disorders) | 4 | 3
Gout (Metabolism and nutrition disorders) | 4 | 3
Hypotension (Vascular disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 5 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Bronchitis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Hypertension (Vascular disorders) | 3 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03759392/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT03759392/SAP_001.pdf